CLINICAL TRIAL: NCT02250937
Title: Allogeneic Transplantation Using Venetoclax, Timed Sequential Busulfan,Cladribine, and Fludarabine Conditioning in Patients With AML and MDS
Brief Title: Venetoclax and Sequential Busulfan, Cladribine, and Fludarabine Phosphate Before Donor Stem Cell Transplant in Treating Patients With Acute Myelogenous Leukemia or Myelodysplastic Syndrome
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0431; NCI-2014-02324 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0431 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-09-24; First posted 2014-09-26 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Stem Cell Transplantation; Busulfan; Cladribine; fludarabine phosphate; Peripheral Blood Stem Cell Transplantation; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (busulfan days -13 and -12 before PBSCT) (Experimental): PREPARATIVE REGIMEN: Patients receive venetoclax PO QD on days -22 to -3 and busulfan IV over 3 hours on days -13 and -12. Patients then receive fludarabine phosphate IV over 1 hour, cladribine IV over 2 hours, and busulfan IV over 3 hours on days -6 to -3.
  TRANSPLANT: Patients undergo allogeneic PBSCT on day 0.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Busulfan; Drug: Cladribine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Pharmacological Study; Drug: Venetoclax
- Arm II (busulfan days -20 and -13 before PBSCT) (Experimental): PREPARATIVE REGIMEN: Patients receive venetoclax PO QD on days -22 to -3 and busulfan IV over 3 hours on days -20 and -13. Patients then receive fludarabine phosphate IV over 1 hour, cladribine IV over 2 hours, and busulfan IV over 3 hours on days -6 to -3.
  TRANSPLANT: Patients undergo allogeneic PBSCT on day 0.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Busulfan; Drug: Cladribine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Pharmacological Study; Drug: Venetoclax

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic PBSCT
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Cladribine — Given IV
  Other Names: 2-CdA; 2CDA; CdA; Cladribina; Leustat; Leustatin; Leustatine; RWJ-26251
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo allogeneic PBSCT
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Other: Pharmacological Study — Correlative studies
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This randomized phase II trial studies how well venetoclax and sequential busulfan, cladribine, and fludarabine phosphate before donor stem cell transplant work in treating patients with acute myelogenous leukemia or myelodysplastic syndrome. Giving chemotherapy before a donor peripheral blood stem cell transplant helps kill cancer cells in the body and helps make room in the patient's bone marrow for new blood-forming cells (stem cells) to grow. When the healthy stem cells from a donor are infused into a patient, they may help the patient's bone marrow make more healthy cells and platelets and may help destroy any remaining cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare progression free survival of two schedules of venetoclax, timed sequential busulfan, cladribine and fludarabine conditioning regimen in patients with acute myelogenous leukemia (AML) and myelodysplastic syndrome (MDS).

SECONDARY OBJECTIVES:

I. Compare overall survival between the two schedules. II. Compare non relapse mortality between the two schedules. III. Compare neutrophil and platelet engraftment between the two schedules. IV. Compare acute and chronic graft-versus-host disease (GVHD) between the two schedules.

V. Compare cumulative incidence of relapse between the two schedules. VI. Compare grade III/IV toxicity between the two schedules.

TERTIARY OBJECTIVES:

I. To study chemotherapy resistance. II. To study deoxyribonucleic acid (DNA) damage. III. To study immune recovery and cytokines (both in plasma and cells). IV. To study BCL-2 family expression, stem cell surface markers and intracellular signaling markers in AML cells at the time of relapse.

OUTLINE:

PREPARATIVE REGIMEN: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive venetoclax orally (PO) once daily (QD) on days -22 to -3 and busulfan intravenously (IV) over 3 hours on days -13 and -12. Patients then receive fludarabine phosphate IV over 1 hour, cladribine IV over 2 hours, and busulfan IV over 3 hours on days -6 to -3.

ARM II: Patients receive venetoclax PO QD on days -22 to -3 and busulfan IV over 3 hours on days -20 and -13. Patients then receive fludarabine phosphate IV over 1 hour, cladribine IV over 2 hours, and busulfan IV over 3 hours on days -6 to -3.

TRANSPLANT: Patients undergo allogeneic peripheral blood stem cell transplant (PBSCT) on day 0.

After completion of study treatment, patients are followed up for 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven acute myeloid leukemia or myelodysplastic syndrome with persistent disease or in remission
* Human leukocyte antigen (HLA)-identical sibling or 8/8 matched unrelated donor transplant
* Patients age 18 to 70 years old; eligibility for pediatric patients will be determined in conjunction with an MD Anderson Cancer Center (MDACC) pediatrician; patients age 2-17 years may be enrolled after at least 10 adults (ages 18-70 years old) have been assessed for safety at day 30
* Direct bilirubin < 1 mg/dl
* Alanine aminotransferase (ALT) < 3 times upper limit of normal
* Creatinine clearance > 50 ml/min (calculated creatinine clearance is permitted)
* Forced expiratory volume in 1 second (FEV1) >= 50% of expected corrected for hemoglobin and/or volume
* Forced vital capacity (FVC) >= 50% of expected corrected for hemoglobin and/or volume
* Diffusing capacity of the lungs for carbon monoxide (DLCO) >= 50% of expected corrected for hemoglobin and/or volume
* Children unable to perform pulmonary function tests (e.g., less than 7 years old) pulse oximetry of >= 92% on room air
* Left ventricular ejection fraction (LVEF) >= 40%
* Patient, legally authorized representative (LAR), or parent able to sign informed consent; able to give assent for patients age 7-17
* Negative beta human chorionic gonadotropin (HCG) test in a woman with child bearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization; women of child bearing potential must be willing to use an effective contraceptive measure while on study
* Performance score of >= 70 by Karnofsky/Lansky or performance status (PS) 0 or 1 (Eastern Cooperative Oncology Group [ECOG] =< 1)

Exclusion Criteria:

* Prior allogeneic or autologous transplantation
* Uncontrolled infections
* Human immunodeficiency virus (HIV) seropositivity
* Hematopoietic cell transplantation (HCT) co-morbidity index score > 3; the principal investigator is the final arbiter of eligibility for comorbidity score > 3
* Patients with prior coronary artery disease

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2014-10-27 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | At 6 months
  The method of Kaplan and Meier will be used to estimate distribution of progression free survival.
Disease free survival (DFS) | Up to 2.5 years
  Will test whether there is strong evidence that DFS differs between the two arms using a stratified log-rank test. Will use the Lan-DeMets alpha spending approach with an O'Brien-Fleming stopping boundary to compare the two arms.

SECONDARY OUTCOMES:
Incidence of toxicity of these regimens | Up to 2.5 years
Cumulative incidence of acute graft versus host disease (GVHD) | Up to 2.5 years
  Will use the method of Gooley et al to estimate the cumulative incidence of acute GVHD. Will use the method of Fine and Gary to fit regression models to the cumulative incidence outcomes.
Cumulative incidence of chronic GVHD | Up to 2.5 years
  Will use the method of Gooley et al to estimate the cumulative incidence of chronic GVHD. Will use the method of Fine and Gary to fit regression models to the cumulative incidence outcomes.
Overall survival | Up to 2.5 years
  The method of Kaplan and Meier will be used to estimate the distribution of overall survival. Cox proportional hazards regression analysis will be used to model the association between overall survival and covariates of interest.
Time to neutrophil engraftment | Up to 2.5 years
  The method of Kaplan and Meier will be used to estimate time to neutrophil engraftment.
Time to platelet engraftment | Up to 2.5 years
  The method of Kaplan and Meier will be used to estimate time to platelet engraftment.
Cumulative incidence of relapse | Up to 2.5 years
  Will use the method of Gooley et al to estimate the cumulative incidence of relapse. Will use the method of Fine and Gary to fit regression models to the cumulative incidence outcomes.
Non-relapse mortality | Up to 2.5 years
  Will use the method of Gooley et al to estimate the cumulative incidence of non-relapse mortality. Will use the method of Fine and Gary to fit regression models to the cumulative incidence outcomes. Logistic regression will be used to model the association between 100-day NRM and clinical and demographic covariates of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Uday R Popat, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org